CLINICAL TRIAL: NCT01191801
Title: A Phase 3, Randomized, Controlled, Double-Blind, Multinational Clinical Study of the Efficacy and Safety of Vosaroxin and Cytarabine Versus Placebo and Cytarabine in Patients With First Relapsed or Refractory Acute Myeloid Leukemia (VALOR)
Brief Title: Study of Vosaroxin or Placebo in Combination With Cytarabine in Patients With First Relapsed or Refractory AML
Acronym: VALOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VOS-AML-301; 2010-021961-61 (EudraCT Number)
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2017-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Leukemia; Acute Myeloid Leukemia; Hematologic; Hematologic diseases; Blood; Cancer; Malignancy; Vosaroxin; Cytarabine; First Relapsed AML; Refractory AML; VALOR; Sunesis; Voreloxin; SNS-595
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Hematologic Diseases; Neoplasms | interventions — vosaroxin; Cytarabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: vosaroxin + cytarabine (Experimental): vosaroxin (short IV infusion within 10 minutes) on days 1 and 4: cytarabine on days 1 through 5; a maximum of 2 cycles of Induction and 2 cycles for Consolidation
  Interventions: Drug: vosaroxin + cytarabine
- Group B: placebo + cytarabine (Placebo Comparator): placebo (short IV infusion within 10 minutes and volume matched to vosaroxin) on days 1 and 4: cytarabine on days 1 through 5; a maximum of 2 cycles of Induction and 2 cycles for Consolidation
  Interventions: Drug: placebo + cytarabine

INTERVENTIONS:
Drug: vosaroxin + cytarabine — Vosaroxin days 1 and 4: 90 mg/m2 for induction 1; 70 mg/m2 for all other cycles
  Cytarabine 1 g/m2 daily on days 1-5 (IDAC)
  Arms: Group A: vosaroxin + cytarabine
Drug: placebo + cytarabine — Placebo days 1 and 4: volume matched to vosaroxin
  Cytarabine 1 g/m2 daily on days 1-5 (IDAC)
  Other Names: control
  Arms: Group B: placebo + cytarabine

SUMMARY:
This study compared treatment groups of patients treated with vosaroxin and cytarabine versus patients treated with placebo and cytarabine.

DETAILED DESCRIPTION:
The study includes additional objectives to ones listed above as Outcome Measures. These additional objectives also compared treatment groups in the following:

CR + CRp rate, defined as CR + CRp based on modified IWG response criteria.

Combined CR rate (CR+CRp+CRi).

Percentage of patients who have post-treatment (subsequent) transplantation.

Percentage of patients who received subsequent non-protocol therapy (including transplantation).

Safety and tolerability.

In keeping with FDA guidance for adaptive trial designs, the study incorporated an independent DSMB (Drug Safety Monitoring Board) to address potential uncertainty concerning the true treatment affect between the treatment groups and to address a deterioration of power from a small difference. Sunesis remained blinded and had no involvement in the interim data analysis, interpretation, or adaptive design. Based on the results of the interim data analysis the DSMB recommended an increase in the target number of deaths from 375 in 450 patients to 562 in 675 patients which based on a 5% dropout rate increased enrollment from 475 to 712.

The primary analysis was performed when the target number of deaths had been achieved based on a permuted block randomization procedure, stratified by disease status (refractory, first relapse with duration of first CR or CRp ≥ 90 days and < 12 months, or first relapse with duration of first CR or CRp ≥ 12 months and ≤ 24 months), age (< 60 years or ≥ 60 years), and geographic location (US or outside US). The study included periods of screening, treatment / hematologic recovery, post-treatment follow-up, and long-term follow-up for survival.

Follow-up was monthly during the first year, every 2 months during the second year, and every 3 months thereafter until death, withdrawal of consent, or loss to follow-up, whichever occurred first. Long-term follow-up began for all patients when the required number of deaths for primary analysis had been met; thereafter, survival data were collected every 4 months until death, withdrawal of consent, or loss to follow-up, whichever occurred first.

The long term follow-up for this study continues at this time and the September 2014 date reflects database lock for primary analyses reflected in the Results Section. During long term follow-up Sunesis is not collecting Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed, written informed consent
* At least 18 years of age
* Had a diagnosis of AML according to World Health Organization (WHO) classification
* First relapsed or refractory AML (refractory to initial induction therapy) with at least 5% blasts by bone marrow or aspirate or 1% blasts in peripheral blood with additional requirements for relapsed or refractory
* Had an ECOG score of 0-2
* Had adequate liver and renal function as indicated by certain laboratory values
* Had adequate cardiac function (left ventricular ejection fraction at least 40% by multiple gated acquisition scan or ECG)
* Nonfertile or agreed to use an adequate method of contraception until 30 days after the last treatment
* Had any clinically significant nonhematologic toxicity after prior chemotherapy recovered to Grade 1 per NCI-CTCAE

Exclusion Criteria:

* Had acute promyelocytic leukemia
* Had more than 2 cycles of induction therapy for AML
* Had completed a single cycle of treatment containing a total dose of 5 g/m2 or more of cytarabine within 90 days before randomization
* Refractory to or relapsed within the previous 3 months after therapy with an IDAC- or HIDAC-containing regimen
* Had received a hematopoietic stem cell transplant (HSCT) within the previous 90 days
* Had received active immunosuppressive therapy for graft-versus-host disease (GVHD) within 2 weeks before study start
* Had any other severe concurrent disease, or have a history of serious disease involving the heart, kidney, liver, or other organ system
* Had evidence of central nervous system involvement of active AML
* Had other active malignancies (including other hematologic malignancies) or been diagnosed with other malignancies within the last 12 months, except nonmelanoma skin cancer or cervical intraepithelial neoplasia
* Had an active, uncontrolled infection
* Had received any other investigational therapy within 14 days or not recovered from acute affects of the other investigational therapy
* Had received prior or current hydroxyurea or medications to reduce blast count within 24 hours before randomization
* Had received previous treatment with vosaroxin
* Pregnant or lactating
* Had any other medical, psychological, or social condition that may interfere with consent, study participation, or follow-up
* Had known HIV seropositivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2010-12-17; Primary Completion 2014-09-26 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Neuman, MD, Study Director — Sunesis Pharmaceuticals
Locations (124):
- United States (38):
  - Moores UCSD Cancer Center, La Jolla, California
  - UCLA Division of Hematology/Oncology, Los Angeles, California
  - Sharp Clinical Oncology Research, San Diego, California
  - University of California San Francisco, San Francisco, California
  - HCA HealthONE - Rocky Mountain Blood and Marrow Transplant Program, Denver, Colorado
  - George Washington University-Medical Faculty Associates, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Georgia Health Sciences University, Augusta, Georgia
  - Rush University Medical Center, Division of Hematology/Oncology, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - St. Francis Medical Group Oncology and Hematology Specialists, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Ellis Fischel Cancer Center, University of Missouri Health Care, Columbia, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - North Shore Long Island Jewish Health System, Lake Success, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - New York Medical College, Division of Oncology/Hematology, Valhalla, New York
  - Mecklenburg Medical Group, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University Hospitals fo Cleveland, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Family Cancer Center, Memphis, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - The University of Texas, M.D. Anderson Cancer Center, Department of Leukemia, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Department of Medicine Section of Hematology/Oncology, West Virginia University Hospitals, Mary Babb Randolph Cancer Center, West Virginia University, Morgantown, West Virginia
- Australia (11):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Haematology Department, Gosford Hospital, Gosford, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Haematology and Bone Marrow Transplant Unit, Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Andrew Love Cancer Center, Geelong Hospital, Barwon Health, Geelong, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Department of Clinical Haematology and BMT Service, Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (4):
  - Universitatsklinik Graz, Universitatsklinik fur Innere Medizin, Abteilung fur Hamatologie, Graz
  - University Hospital for Internal Medicine V, Innsbruck Medical University, Innsbruck
  - Landeskrankenhaus Salzburg, Universitaetsklinik fur innere Medizin lll, Universitaetsklinikum der PMU, Salzburg
  - AKH Wien / MedUniWien Universtatsklinik fur Innere Medizin 1, Vienna
- Belgium (6):
  - ZNA Middleheim Lindendreef 1, Antwerp
  - ZNA Stuivenberg, Lange Beeldekensstraat 267, Antwerp
  - AZ St.-Jan Brugge-Oostende AV, Bruges
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Leuven, campus Gasthuisberg, Department of Haematology, Leuven
  - H.-Hartziekenhuis Roeselare - Menen vzw, Roeselare
- Canada (5):
  - Division of Hematology, Vancouver General Hospital, Vancouver, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - University Health Network, Princess Margaret Hospital, Toronto, Ontario
  - Charles LeMoyne Hospital, Greenfield Park, Quebec
- Czechia (3):
  - Fakultni nemocnice Kralovske Vinohrady, Oddeleni klinicke hematologie, Prague, Srobarova
  - Fakultni nemocnice Brno, Interni hematoonkologicka klinika, Brno
  - Fakultni nemocnice Hradec Kralove, 2. Interni klinika-oddeleni klinicke hematologie, Hradec Králové
- France (9):
  - CHU Lille, Service des maladies du sang, Hopital Huriez, Lille, Lille Cedex
  - CHU Angers, Service des maladies du sang, Angers
  - Hopital Avicenne- Departement Onco-hematologie, Bobigny
  - Hopital Mignot, Le Chesnay
  - Institut Paoli Calmettes, Marseille
  - CHU Nantes Hotel Dieu, Service d'hematologie clinique, Nantes
  - CHU de Bordeaux- Hopital Haut-Leveque, Centre Francois Magendle, Pessac
  - Centre Hospitalier Lyon Sud - Service d'Hematologie - Pavillon Marcel Berard - Bat. 1G - 1er etage, 165 Chemin du grand Revoyet, Pierre-Bénite
  - Service d'hematologie- Hopital Purpan- CHU de Toulouse, Toulouse
- Germany (9):
  - St. Johannes-Hospital, Duisburg
  - Klinikum Frankfurt am Main-Hochst, Department of Hematology and Oncology, Klinikum Frankfurt Academic Hospital of the University of Frankfurt, Frankfurt
  - Universitatsklinikum Hamburg-Eppendorf; ll. Medizinische Klinik und Poliklinik; Onkologie, Hamatologie und Knochenmarktransplantation, Hamburg
  - Medizinische Hochschule Hannover, Abteilung Hamatologie, Hanover
  - SLK-Kliniken Heilbronn GmbH, Medizinische Klinik, Heilbronn
  - Staedtisches Krankenhaus Kiel GmbH, Infektionsambulanz der 2. Medizinischen Klinik, Kiel
  - Klinikum St. Georg gGmbH; Klinik fur Internistische Onkologie/Hamatologie, Leipzig
  - Klinikum rechts der Isar der Technischen Universitat Munchen lll, Medizinische Klinik, Munich
  - University Hospital of Muenster, Münster
- Hungary (4):
  - University of Debrecen Medical and Health Sciences Center, Debrecen
  - Petz Aladar County Hospital, Győr
  - kaposi Mor Oktato Korhaz Belgyogyaszati Osztaly, Kaposvár
  - Szegedi Tudomanyegyetem, 11. Belgyogyaszati Klinika, Szeged
- Italy (7):
  - Ospedale "A. Perrino", U.O. Compessa di Ematologia, Brindisi
  - Azienda Ospedaliero-Universitaria Sant'Anna, Sezione di Ematologia, Dipartmento di Science Biomediche e Terapie Avanzate, Ferrara
  - Ospedaliera Universitaria San Martino di Genova, Genova
  - Ospedale "Vito Fazzi", U.O Ematologia, Lecce
  - AORN "A. Cardarelli", U.O.S.C. Ematologia con TMO, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore Della Carita, Struttura Complessa Direzione Universitaria Ematologia, Novara
  - Fondazione IRCCS, Policlinico S. Matteo - Dipartimento di Ematologia, Pavia
- New Zealand (4):
  - Haematology Research, Auckland District Health Board, Auckland City Hospital, Grafton, Auckland
  - Canterbury Health Laboratories, Christchurch
  - Department of Haematology, Waikato Hospital, Hamilton
  - Regional Cancer Treatment Service, Palmerston North Hospital, Palmerston North
- Poland (3):
  - Uniwersyteckle Centrum Kliniczne, Gdansk
  - Klinika Hematologii i Chorob Rozrostowych Ukladu Krwiotworczego, Szpital Kliniczny Przemiemienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Division of Hematology-Oncology, Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Dept. of Hematology, Asan Medical Center, Seoul
- Spain (9):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital del Mar, Barcelona
  - Centro Oncologico MD Anderson International Espana, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Sont Llatzer, Palma de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitari Politecnic la Fe Hematology Department, Valencia
- United Kingdom (8):
  - Blackpool Victoria Hospital, Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital, Cambridge
  - Department of Haematology, University Hospital of Wales, Cardiff
  - Queen's Centre for Oncology and Hematology, Castle Hill Hospital, Cottingham
  - Leicester Royal Infirmary, University Hospitals of Leicester, NHS Trust, Leicester
  - Department of Haematology, Royal Liverpool University Hospital, Liverpool
  - Department of Haematology, Guy's Hospital, London
  - Central Manchester University Hospitals NHS Trust, Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: Yes
De-identified data of individual participants experiencing Serious Adverse Events

REFERENCES:
- [Derived] Ravandi F, Ritchie EK, Sayar H, Lancet JE, Craig MD, Vey N, Strickland SA, Schiller GJ, Jabbour E, Erba HP, Pigneux A, Horst HA, Recher C, Klimek VM, Cortes J, Roboz GJ, Odenike O, Thomas X, Havelange V, Maertens J, Derigs HG, Heuser M, Damon L, Powell BL, Gaidano G, Carella AM, Wei A, Hogge D, Craig AR, Fox JA, Ward R, Smith JA, Acton G, Mehta C, Stuart RK, Kantarjian HM. Vosaroxin plus cytarabine versus placebo plus cytarabine in patients with first relapsed or refractory acute myeloid leukaemia (VALOR): a randomised, controlled, double-blind, multinational, phase 3 study. Lancet Oncol. 2015 Sep;16(9):1025-1036. doi: 10.1016/S1470-2045(15)00201-6. Epub 2015 Jul 30. PMID 26234174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 320 patients enrolled in 30 US sites:391 patients enrolled at 71 sites outside of the US (Canada, Europe, Australia, New Zealand, and Republic of Korea)
Pre-assignment Details: Six patients were randomized but never received treatment due to death prior to beginning treatment: 4 assigned to receive vosaroxin/cytarabine; 2 assigned to receive placebo/cytarabine.
Groups:
- Group A (Vosaroxin/Cytarabine): Vosaroxin on Days 1 and 4 (90 mg/m2 induction 1; 70 mg/m2 all other cycles); cytarabine 1 g/m2 daily on Days 1 through 5
- Group B (Placebo/Cytarabine): Placebo (volume matched to vosaroxin) on Days 1 and 4; cytarabine 1 g/m2 daily on Days 1 through 5
Period: Overall Study
Arm/Group | Group A (Vosaroxin/Cytarabine) | Group B (Placebo/Cytarabine)
Started | 356 | 355
Completed | 40 | 18
Not Completed | 316 | 337
Not completed — Death | 36 | 12
Not completed — Lack of Efficacy | 176 | 258
Not completed — Adverse Event | 9 | 8
Not completed — Protocol Violation | 2 | 4
Not completed — Physician Decision | 47 | 24
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Not Provided | 45 | 27

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population: Patients who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Vosaroxin/Cytarabine) | Group B (Placebo/Cytarabine) | Total
Number analyzed (Participants) | 356 | 355 | 711
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11.51) | 60.2 (12.49) | 60.6 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 163 | 317
  Male | 202 | 192 | 394
Region of Enrollment [Number; unit: participants]
  Hungary | 8 | 11 | 19
  United States | 161 | 159 | 320
  United Kingdom | 15 | 10 | 25
  Spain | 9 | 8 | 17
  New Zealand | 4 | 3 | 7
  Canada | 10 | 10 | 20
  Czech Republic | 5 | 6 | 11
  Austria | 4 | 4 | 8
  Belgium | 17 | 19 | 36
  Poland | 3 | 1 | 4
  Korea, Republic of | 10 | 5 | 15
  Italy | 20 | 18 | 38
  Australia | 25 | 20 | 45
  France | 38 | 50 | 88
  Germany | 27 | 31 | 58

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Vosaroxin + cytarabine patient survival versus placebo + cytarabine patient survival
Time Frame: Up to 5 years or duration of study
Population: The intent-to-treat (ITT) population which consists of all patients enrolled (randomly assigned to treatment group).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A (Vosaroxin/Cytarabine) | Group B (Placebo/Cytarabine)
Number analyzed (Participants) | 356 | 355
Months | 7.5 [6.4 to 8.5] | 6.1 [5.2 to 7.1]
Statistical Analysis 1: Comparison: Group A (Vosaroxin/Cytarabine) vs Group B (Placebo/Cytarabine); Test type: Superiority or Other; p = 0.0305, Unstratified Log Rank — Unstratified one sided P-Value; Since the sample size was increased, the primary analysis used the weighted statistic proposed by Cui, Hung, and Wang (Cui 1999); Cox Proportional Hazard = 0.87

2. Secondary Outcome: Complete Remission (CR) Rate Based on Modified International Working Group (IWG) Criteria.
Description: Group A (Vosaroxin + cytarabine) patient CR as compared to Group B (placebo + cytarabine) patient CR. Complete remission (CR) is typically defined using IWG criteria as bone marrow blast count of less than 5% with adequate recovery of peripheral blood counts.
Time Frame: Up to 5 years or duration of study
Population: The percentage of patients who achieved CR was adjudicated by the CPARR (Central Pathology and Response Review) panel using modified IWG response criteria. The outcome measure reflects the Intent to Treat Population.
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Group A (Vosaroxin/Cytarabine) | Group B (Placebo/Cytarabine)
Number analyzed (Participants) | 356 | 355
percentage of particpants | 30.1 [25.3 to 35.1] | 16.3 [12.6 to 20.6]
Statistical Analysis 1: Comparison: Group A (Vosaroxin/Cytarabine) vs Group B (Placebo/Cytarabine); Test type: Superiority or Other; p < 0.0001, Chi-squared — Two sided P-Value

3. Secondary Outcome: All Cause Mortality
Description: Vosaroxin + cytarabine mortality versus placebo + cytarabine mortality
Time Frame: 30 Days
Population: Safety Population (705)
Measure: Number (95% Confidence Interval); unit: percentage of Participants in the Group
Arm/Group | Group A (Vosaroxin/Cytarabine) | Group B (Placebo/Cytarabine)
Number analyzed (Participants) | 355 | 350
percentage of Participants in the Group | 7.9 [5.3 to 11.2] | 6.6 [4.2 to 9.7]

4. Secondary Outcome: All Cause Mortality
Description: Vosaroxin + cytarabine mortality versus placebo + cytarabine mortality
Time Frame: 60 Days
Population: Safety Population (705)
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group A (Vosaroxin/Cytarabine) | Group B (Placebo/Cytarabine)
Number analyzed (Participants) | 355 | 350
percentage of Participants | 19.7 [15.7 to 24.2] | 19.4 [15.4 to 24.0]

5. Other Pre Specified Outcome: Overall Remission (OR) Rate Based on the IWG Response Criteria
Description: Group A patient OR compared to Group B patient OR
  Overall Remission includes Complete Remission (CR), Complete Remission with incomplete platelet recovery (CRp), Complete Remission with incomplete blood count recovery (CRi), and Partial Remission (PR). Complete remission means bone marrow blast count of less than 5% with adequate recovery of peripheral blood counts as typically defined by the IWG. Both CRi and CRp refer complete remission but with incomplete blood count and platelet recovery, respectively. PR, or partial remission, refers to remission in which bone marrow contains blast counts between 5 and 25 percent.
Time Frame: Up to 5 years or the duration of the study
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A (Vosaroxin/Cytarabine) | Group B (Placebo/Cytarabine)
Number analyzed (Participants) | 356 | 355
percentage of participants | 37.9 [32.9 to 43.2] | 18.9 [14.9 to 23.3]
Statistical Analysis 1: Comparison: Group A (Vosaroxin/Cytarabine) vs Group B (Placebo/Cytarabine); Test type: Superiority or Other; p < 0.0001, Chi-squared — Two sided P-Value

6. Other Pre Specified Outcome: Event Free Survival (EFS)
Time Frame: Up to 5 years or duration of study
Population: Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A (Vosaroxin/Cytarabine) | Group B (Placebo/Cytarabine)
Number analyzed (Participants) | 356 | 355
months | 1.9 [1.6 to 2.2] | 1.3 [1.2 to 1.4]
Statistical Analysis 1: Comparison: Group A (Vosaroxin/Cytarabine) vs Group B (Placebo/Cytarabine); Test type: Superiority or Other; p < 0.0001, Log Rank — Unstratified one-sided P-Value; Hazard Ratio (HR) = 0.67

7. Other Pre Specified Outcome: Leukemia-Free Survival (LFS)
Description: Durability of remission (CR) assessed by LFS
Time Frame: Up to 5 years or the duration of the study
Population: Subset of Intent to Treat patients that have a Measured CR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A (Vosaroxin/Cytarabine) | Group B (Placebo/Cytarabine)
Number analyzed (Participants) | 107 | 58
Months | 11 [8.3 to 14.3] | 8.7 [6.5 to 18.0]
Statistical Analysis 1: Comparison: Group A (Vosaroxin/Cytarabine) vs Group B (Placebo/Cytarabine); Test type: Superiority or Other; p = 0.3134, Log Rank — One sided P-Value; Hazard Ratio (HR) = 0.89

ADVERSE EVENTS:
Time Frame: Adverse Event reported below reflects time from first patient randomization 17 December 2010 to database lock for primary analysis 26 September 2014. The Tables show Incidence of Treatment Emergent Adverse Events.
Arm/Group | Group A (Vosaroxin/Cytarabine) | Group B (Placebo/Cytarabine)
All-Cause Mortality (participants affected / at risk) | 273/355 | 288/350
Serious Adverse Events (participants affected / at risk) | 197/355 | 125/350
Other Adverse Events (participants affected / at risk) | 354/355 | 349/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Vosaroxin/Cytarabine) (N=355) | Group B (Placebo/Cytarabine) (N=350)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 40 | 26
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Pure white cell aplasia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Myopericarditis (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Diabetes insipidus (Endocrine disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Caecitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Ileitis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Neutropenic colitis (Gastrointestinal disorders) | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 3 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 12 | 5
Asthenia (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 0 | 1
Medical device complication (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 3
Sudden death (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Abscess neck (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 2
Anorectal cellulitis (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1
Aspergilloma (Infections and infestations) | 1 | 0
Aspergillosis (Infections and infestations) | 2 | 1
Bacteraemia (Infections and infestations) | 30 | 10
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 4 | 1
Clostridial infection (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Enterobacter infection (Infections and infestations) | 1 | 0
Enterobacter sepsis (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 2 | 0
Enterocolitis bacterial (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 1
Escherichia sepsis (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fungaemia (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 2 | 2
Fungal sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Infusion site cellulitis (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 9 | 7
Perirectal abscess (Infections and infestations) | 3 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 27 | 17
Pneumonia fungal (Infections and infestations) | 7 | 2
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 1
Pseudomonas infection (Infections and infestations) | 1 | 2
Pulmonary mycosis (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 31 | 15
Septic embolus (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 7 | 6
Sinusitis (Infections and infestations) | 0 | 1
Sinusitis aspergillus (Infections and infestations) | 0 | 1
Sinusitis fungal (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 2
Staphylococcal infection (Infections and infestations) | 4 | 1
Streptococcal bacteraemia (Infections and infestations) | 3 | 0
Systemic candida (Infections and infestations) | 1 | 2
Thrombophlebitis septic (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 4
Urinary tract infection enterococcal (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0
Viral pericarditis (Infections and infestations) | 1 | 0
Vulval abscess (Infections and infestations) | 1 | 0
Vulval cellulitis (Infections and infestations) | 0 | 1
Vulvovaginitis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2
Neurotoxicity (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 2 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism arterial (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 2 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Vosaroxin/Cytarabine) (N=355) | Group B (Placebo/Cytarabine) (N=350)
Anaemia (Blood and lymphatic system disorders) | 95 | 104
Febrile neutropenia (Blood and lymphatic system disorders) | 143 | 97
Neutropenia (Blood and lymphatic system disorders) | 70 | 50
Thrombocytopenia (Blood and lymphatic system disorders) | 88 | 90
Atrial fibrillation (Cardiac disorders) | 22 | 16
Tachycardia (Cardiac disorders) | 32 | 29
Abdominal distension (Gastrointestinal disorders) | 20 | 10
Abdominal pain (Gastrointestinal disorders) | 79 | 46
Abdominal pain upper (Gastrointestinal disorders) | 31 | 33
Constipation (Gastrointestinal disorders) | 136 | 141
Diarrhoea (Gastrointestinal disorders) | 243 | 121
Dry mouth (Gastrointestinal disorders) | 22 | 12
Dyspepsia (Gastrointestinal disorders) | 46 | 17
Dysphagia (Gastrointestinal disorders) | 20 | 7
Haemorrhoids (Gastrointestinal disorders) | 30 | 14
Nausea (Gastrointestinal disorders) | 218 | 167
Oral pain (Gastrointestinal disorders) | 21 | 6
Stomatitis (Gastrointestinal disorders) | 169 | 64
Vomiting (Gastrointestinal disorders) | 135 | 73
Asthenia (General disorders) | 60 | 43
Chest pain (General disorders) | 29 | 19
Chills (General disorders) | 61 | 46
Fatigue (General disorders) | 107 | 94
Oedema peripheral (General disorders) | 96 | 69
Pain (General disorders) | 21 | 32
Pyrexia (General disorders) | 118 | 106
Bacteraemia (Infections and infestations) | 18 | 6
Oral candidiasis (Infections and infestations) | 18 | 16
Oral herpes (Infections and infestations) | 23 | 4
Pneumonia (Infections and infestations) | 22 | 19
Procedural pain (Injury, poisoning and procedural complications) | 8 | 20
Transfusion reaction (Injury, poisoning and procedural complications) | 18 | 16
Alanine aminotransferase increased (Investigations) | 29 | 17
Aspartate aminotransferase increased (Investigations) | 24 | 16
Blood creatinine increased (Investigations) | 18 | 10
Platelet count decreased (Investigations) | 23 | 29
White blood cell count decreased (Investigations) | 24 | 21
Decreased appetite (Metabolism and nutrition disorders) | 126 | 59
Fluid overload (Metabolism and nutrition disorders) | 18 | 16
Fluid retention (Metabolism and nutrition disorders) | 19 | 23
Hyperglycaemia (Metabolism and nutrition disorders) | 43 | 33
Hypoalbuminaemia (Metabolism and nutrition disorders) | 30 | 20
Hypocalcaemia (Metabolism and nutrition disorders) | 49 | 25
Hypokalaemia (Metabolism and nutrition disorders) | 170 | 102
Hypomagnesaemia (Metabolism and nutrition disorders) | 95 | 58
Hyponatraemia (Metabolism and nutrition disorders) | 31 | 20
Hypophosphataemia (Metabolism and nutrition disorders) | 56 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 38
Bone pain (Musculoskeletal and connective tissue disorders) | 21 | 18
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 34 | 44
Dizziness (Nervous system disorders) | 32 | 35
Dysgeusia (Nervous system disorders) | 25 | 7
Headache (Nervous system disorders) | 103 | 93
Anxiety (Psychiatric disorders) | 43 | 56
Confusional state (Psychiatric disorders) | 25 | 19
Depression (Psychiatric disorders) | 30 | 22
Insomnia (Psychiatric disorders) | 78 | 70
Cough (Respiratory, thoracic and mediastinal disorders) | 71 | 44
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 63 | 44
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 56 | 55
Hiccups (Respiratory, thoracic and mediastinal disorders) | 23 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 46 | 41
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 26 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 9
Erythema (Skin and subcutaneous tissue disorders) | 25 | 16
Petechiae (Skin and subcutaneous tissue disorders) | 27 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 41 | 28
Rash (Skin and subcutaneous tissue disorders) | 53 | 37
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 | 10
Hypertension (Vascular disorders) | 40 | 32
Hypotension (Vascular disorders) | 66 | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days